CLINICAL TRIAL: NCT01567176
Title: Circulating Expression Measurement of a Sirtuin Protein Isoform, Sirt6, as an Early Marker of Aging Quality
Brief Title: Circulating SIRT6 Expression, Effect on Aging Quality
Acronym: Sirt6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011.674
Record Dates: First submitted 2012-03-08; First posted 2012-03-30 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2012-02

CONDITIONS: Aging
Keywords: Sirtuins; Aging; Metabolic disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — It is a single cross sectional study. All outcome measures will be taken during the investigation with physical examination, questionnaire and a blood sample

SUMMARY:
This study follows the results of the COMPALICLAMP study (NCT00951392) where the investigators showed a differential expression of sirtuins protein isoforms, Sirt6, in muscle depending on the quality of aging. The investigators seek to confirm this difference in expression level of circulating leukocytes on a larger sample.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers from the SUVIMAX 2 aging cohort
* Men and women
* Older than 60
* Subject with a global aging quality score of 1 or 3 in the SU.VI.MAX. 2 study
* Covered by Health Insurance System

Exclusion Criteria:

* Subject not in compliance with the recommendation of French National Law

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Sirt6 expression in circulating leukocytes based on the aging quality | participants will be followed for the duration of the visit, an expected average of 1 day
  analysis by quantitative RT-PCR method

SECONDARY OUTCOMES:
hand and forearm muscular strength measurement | participants will be followed for the duration of the visit, an expected average of 1 day
  Hand Grip strength test
Physical examination and anthropometric measurement | participants will be followed for the duration of the visit, an expected average of 1 day
  Measurement of the weight, height, waist, hips, blood pressure, pulse.
Cognitive assessment | participants will be followed for the duration of the visit, an expected average of 1 day
  MMSE (Mini Mental State Examination), Five-word test, clock drawing
Physical Activity questionnaire | participants will be followed for the duration of the visit, an expected average of 1 day
  MAQ (Modifiable Activity Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, Pr, Principal Investigator — Centre de recherche en nutrition humaine Rhone-Alpes
Locations (2):
- France (2):
  - Centre de recherche en nutrition humaine Rhone-Alpes, Pierre-Bénite
  - Centre de Recherche en Nutrition Humaine, Pierre-Bénite

REFERENCES:
- [Result] Betry C, Meugnier E, Pflieger M, Grenet G, Hercberg S, Galan P, Kesse-Guyot E, Vidal H, Laville M. High expression of CPT1b in skeletal muscle in metabolically healthy older subjects. Diabetes Metab. 2019 Apr;45(2):152-159. doi: 10.1016/j.diabet.2018.01.018. Epub 2018 Feb 12. PMID 29657112